CLINICAL TRIAL: NCT03240900
Title: Electrical Stimulation for Improving Postoperative Breast Sensation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Estim Breast
Record Dates: First submitted 2017-07-11; First posted 2017-08-07 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Mammaplasty
MeSH Terms: interventions — Electric Stimulation

STUDY DESIGN:
Intervention Model Description: Patients will receive the intervention to one breast and not the other, therefore acting as their own internal control. The laterality of the intervention will be randomized by a coin flip.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only the surgeon will be aware of the laterality of the intervention. The patient will not be performed. All outcomes will be assessed by the investigators, who will be masked to the laterality until the completion of the study when the surgeon will unmask.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Electrical Stimulation Breast (Experimental): Breast that will receive 1 hour of intraoperative electrical stimulation
  Interventions: Device: Electrical Stimulation
- No Electrical Stimulation Breast (Placebo Comparator): The contralateral breast of the patient will receive no electrical stimulation
  Interventions: Procedure: Placebo

INTERVENTIONS:
Device: Electrical Stimulation — Electrical stimulation - a needle attached to an cathode polarity will be placed within the intercostal space near the 4th intercostal nerve. A second needle attached to the anode polarity will be inserted into the serratus anterior muscle. Both electrodes will then be attached to a Grass SD9 stimulator and the voltage and frequency of the stimulation will be titrated to the point where contraction of the intercostal muscles is palpable. It will be maintained at this level for one hour at which point the wires will be removed. This technique is part of the standard of care for peripheral nerve surgeries of the extremities and is proven to be safe in humans.
  Arms: Electrical Stimulation Breast
Procedure: Placebo — This breast will receive no electrical stimulation; the mastectomy and reconstruction will proceed with no intervention.
  Arms: No Electrical Stimulation Breast

SUMMARY:
Described as the "Angelina Jolie Effect", rates of prophylactic mastectomy with immediate implant-based reconstruction are increasing dramatically as more women with genetic predisposition towards breast cancer are seeking surgical prevention. Advances in surgical techniques allow for the creation of an aesthetically pleasing postoperative breast mound; however, a common complaint is the lack of sensation to the skin and nipple of the reconstructed breast due to injury and stretch of the sensory nerves. Numbness of the breast, nipple, and areola is an unnatural feeling for the patient, as well as a potential risk for injury or burns as the woman is unable to feel pain.

Our laboratory has previously shown that electrical stimulation (ES) is an effective way of improving nerve regeneration after injury to the nerves of the upper and lower extremities. Proven to improve motor outcomes following carpal and cubital tunnel release and sensation following injury to the digital nerves, this technique is a likely mechanism of restoring sensation of the breast as well.

In this study, we will follow thirty women undergoing prophylactic skin-sparing mastectomy with immediate implant-based reconstruction. At the time of surgery, patients will be randomly assigned ES to either the right or left breast. That breast will be reconstructed first and stimulated for one hour while the other breast is reconstructed. At the completion of the case, all wires will be removed. We will test sensation (tactile, temperature, 2-point discrimination, sharp/dull discrimination, and protective sensation) prior to surgery then again at 6, 12, 18, and 24 months following surgery to evaluate the effects of ES on sensory return. Patients will be provided with a survey to assess return of erogenous sensation.

DETAILED DESCRIPTION:
Objective: To determine whether intraoperative electrical stimulation enhances sensory recovery following mastectomy with immediate implant reconstruction

Background: There is an increasing trend towards prophylactic mastectomy with immediate implant-based reconstruction for women with genetics predisposing to breast cancer (BRCA-1 and -2). Novel techniques such as fat grafting and nipple creation/tattooing have contributing towards creating an aesthetically pleasing breast mound; however, the majority of women experience non-recoverable significant sensory loss secondary to damage and stretch of the intercostal nerves that provide sensation to the skin, areola, and nipple. Most women will recover minimal sensation around the perimeter of the breast, indicating a potential for sensory return; however, particularly the nipple usually remains numb. An insensate breast feels unnatural to the woman and predisposes her to injury and burns of the reconstruction, which can require additional surgery or cause significant scarring.

Our laboratory has previously shown that electrical stimulation (ES) is safe and significantly improves postoperative outcomes in peripheral nerve injury in animal and human models. ES has been shown to improve return of median and ulnar nerve function following carpal and cubital tunnel release respectively, with improved motor outcomes. Sensory return following digital nerve laceration repair similarly is improved with immediate postoperative ES for one hour.

Methods: Thirty patients that will be undergoing bilateral prophylactic skin-sparing mastectomy with immediate implant-based breast reconstruction will be identified from the practice of two plastic surgeons. Preoperatively, women will be undergo sensory testing to the 4 quadrants of both breasts and the nipples, including testing for tactile sensation, cool detection, 2-point discrimination, heat-pain detection threshold, and sharp-blunt discrimination. A custom-made survey to evaluate erogenous sensation will be completed by the patient, as well as the validated BREAST-Q.

The day of surgery the patient will be randomized to right or left breast for stimulation. Following the mastectomy, the breast to be stimulated will be reconstructed with an implant first in the typical fashion. A percutaneous needle will be passed into the intercostal space alongside the 4th intercostal nerve, and a second needle will be inserted into the serratus anterior muscle . These needles will be attached to the anode and cathode respectively of our electrical stimulator, and the patient will receive 1 hour of intraoperative stimulation titrated to palpable contraction of the intercostal muscle. During this hour, the second breast will undergo reconstruction with no electrical stimulation. At the completion of the hour, the skin will be closed in the normal fashion. The laterality will be blinded to the patient as well as to the investigator who will perform all sensory testing.

Postoperatively, the patient will be evaluated at 1 week, 6 months, 12 months, 18 months and 24 months with the same sensory testing as described previously. Patients will serve as their own internal control, and the sensation of the right vs. left breast will be compared. At the completion of all 2-year evaluations, the study will be unblinded and the stimulated vs. non-stimulated breast outcomes will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Woman aged 18-60 undergoing bilateral, prophylactic nipple/skin-sparing mastectomy with immediate implant reconstruction

Exclusion Criteria:

* Smokers
* Preexisting peripheral neuropathy
* Prior breast surgery

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women undergoing prophylactic bilateral skin/nipple-sparing mastectomy with immediate implant-based breast reconstruction
Enrollment: 30 (Estimated)
Dates: Start 2027-09-01 (Estimated); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Sensation | 12 months
  sensory testing to the 4 quadrants of both breasts and the nipples, including testing for tactile sensation, cool detection, 2-point discrimination, heat-pain detection threshold, and sharp-blunt discrimination

SECONDARY OUTCOMES:
Patient Satisfaction | 12 months
  BREAST-Q Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ming Chan, Principal Investigator — Professor University of Alberta
Locations (2):
- Canada (2):
  - University of Alberta Hospital, Edmonton, Alberta
  - Misericordia Hospital, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No
IPD will be only used by the research team for this study. It will not be shared to other researchers.

REFERENCES:
- [Background] Gahm J, Hansson P, Brandberg Y, Wickman M. Breast sensibility after bilateral risk-reducing mastectomy and immediate breast reconstruction: a prospective study. J Plast Reconstr Aesthet Surg. 2013 Nov;66(11):1521-7. doi: 10.1016/j.bjps.2013.06.054. Epub 2013 Aug 13. PMID 23953096
- [Background] Passavanti MB, Pace MC, Barbarisi A, D'Andrea F, Grella E, Nicoletti GF, Aurilio C. Pain and sensory dysfunction after breast cancer surgery: neurometer CPT evaluation. Anticancer Res. 2006 Sep-Oct;26(5B):3839-44. PMID 17094410
- [Background] Chan KM, Curran MW, Gordon T. The use of brief post-surgical low frequency electrical stimulation to enhance nerve regeneration in clinical practice. J Physiol. 2016 Jul 1;594(13):3553-9. doi: 10.1113/JP270892. Epub 2016 Mar 24. PMID 26864594
- [Background] Gordon T, Brushart TM, Chan KM. Augmenting nerve regeneration with electrical stimulation. Neurol Res. 2008 Dec;30(10):1012-22. doi: 10.1179/174313208X362488. PMID 19079975
- [Background] Gordon T, Amirjani N, Edwards DC, Chan KM. Brief post-surgical electrical stimulation accelerates axon regeneration and muscle reinnervation without affecting the functional measures in carpal tunnel syndrome patients. Exp Neurol. 2010 May;223(1):192-202. doi: 10.1016/j.expneurol.2009.09.020. Epub 2009 Oct 1. PMID 19800329
- [Background] Chan KM, Gordon T, Zochodne DW, Power HA. Improving peripheral nerve regeneration: from molecular mechanisms to potential therapeutic targets. Exp Neurol. 2014 Nov;261:826-35. doi: 10.1016/j.expneurol.2014.09.006. Epub 2014 Sep 16. PMID 25220611
- [Background] Dossett LA, Lowe J, Sun W, Lee MC, Smith PD, Jacobsen PB, Laronga C. Prospective evaluation of skin and nipple-areola sensation and patient satisfaction after nipple-sparing mastectomy. J Surg Oncol. 2016 Jul;114(1):11-6. doi: 10.1002/jso.24264. Epub 2016 Apr 18. PMID 27087574
- [Result] Wong JN, Olson JL, Morhart MJ, Chan KM. Electrical stimulation enhances sensory recovery: a randomized controlled trial. Ann Neurol. 2015 Jun;77(6):996-1006. doi: 10.1002/ana.24397. Epub 2015 May 4. PMID 25727139